CLINICAL TRIAL: NCT03033927
Title: Circulating Tumor Cell and Tumor Tissue Models for Predicting Effective Pancreatic Cancer Response
Brief Title: Predicting Effective Therapy in Pancreatic Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 17-042
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Cancer; Pancreatic Adenocarcinoma
Keywords: Stage IV Pancreatic Cancer; FOLFIRINOX; gem/nab-P chemotherapy; 17-042
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sodium heparin tube collections will be performed at baseline, at each restaging CT scan and at time of first disease progression. K3-EDTA tubes will be collected at baseline and at disease progression.
  In patients who are planning an EGD for the purpose of obtaining a tumor biopsy, portal vein sampling will be offered. Under EUS guidance, a 19-gauge EUS fine needle will be advanced transhepatically into the portal vein and as many as four 7.5 mL K3-EDTA samples of blood will be aspirated, as previously described. Research biopsy will be performed at baseline and, if feasible, at disease progression.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Stage IV Pancreatic Cancer
  Interventions: Diagnostic Test: CTC isolocation and analysis

INTERVENTIONS:
Diagnostic Test: CTC isolocation and analysis — Circulating tumorigenic cell (CTC) isolation and enrichment will be performed using a proprietary invasion assay.

SUMMARY:
The purpose of this phase II study is to develop a test to predict response of pancreatic cancer to different chemotherapy regimens.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of pancreatic adenocarcinoma, confirmed at MSKCC, AJCC stage IV disease at time of enrollment.
* Patient planning to receive treatment with FOLFIRINOX or gem/nab-P chemotherapy, with or without investigational agents.
* Prior surgery, chemotherapy and/or radiation therapy for AJCC Stage I-III pancreatic adenocarcinoma is permitted.
* ECOG performance status 0-2.
* A minimum age of 18 years old.

Exclusion Criteria:

* Prior chemotherapy for AJCC stage IV pancreatic adenocarcinoma
* Known to be HIV positive on antiretroviral therapy
* Prior organ allograft
* Any medical or psychiatric condition that may interfere with the ability to comply with protocol procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced pancreatic adenocarcinoma.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2026-01-24 (Estimated); Study Completion 2026-01-24 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 36 months
  in patients receiving frontline therapy predicted to be effective versus ineffective based on CTC PGx analysis

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Memorial Sloan Kettering Cancer Center Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- [Derived] Yu KH, Park J, Mittal A, Abou-Alfa GK, El Dika I, Epstein AS, Ilson DH, Kelsen DP, Ku GY, Li J, Park W, Varghese AM, Chou JF, Capanu M, Cooper B, Bartlett A, McCarthy D, Sangar V, McCarthy B, O'Reilly EM. Circulating tumor and invasive cell expression profiling predicts effective therapy in pancreatic cancer. Cancer. 2022 Aug 1;128(15):2958-2966. doi: 10.1002/cncr.34269. Epub 2022 Jun 1. PMID 35647938
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org